CLINICAL TRIAL: NCT00507468
Title: Autologous Bone Marrow Transplanted Via Transendocardial Catheter to Chronic Myocardial Infarct Border Zone
Acronym: TABMMI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCardia, Inc. (Industry)
Responsible Party: Peter Altman, BioCardia, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: ABM-MI-10
Record Dates: First submitted 2007-07-22; First posted 2007-07-26 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-11

CONDITIONS: Ventricular Dysfunction; Myocardial Infarction
Keywords: bone marrow; autologous; ejection fraction; left ventricle; heart attack; myocardial infarction; left ventricular dysfunction post myocardial infarction
MeSH Terms: conditions — Ventricular Dysfunction; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Transendocaridal Transplantation of Autologous Bone Marrow — Single treatment, harvest and transplant of patients own bone marrow. Cells are delivered to the myocardium via transendocardial delivery catheter.

SUMMARY:
The object of this open-labeled, uncontrolled pilot study was to investigate the safety and feasibility of percutaneously transplanting autologous bone marrow (ABM) cells into the myocardium using the helical needle transendocardial (TE) delivery system in stable coronary patients with ventricular dysfunction due to chronic myocardial infarction (MI).

A secondary goal was to assess the possibility that such cell injections could improve ejection fraction (EF).

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Able to give informed consent
* Must have documentation of prior myocardial infarction with left ventricular ejection fraction of less than 40 percent at baseline
* Must be a candidate for percutaneous heart catheterization
* Must have identifiable area of transmural scar within the left ventricle

Exclusion Criteria:

* Be a candidate for concurrent ventricular surgical restoration, AICD placement or valvular surgery
* Clinical evidence of infection
* Other complicating cardiovascular abnormalities
* Clinically significant electrocardiographic abnormalities
* Active malignancy
* Recent history or drug or alcohol abuse
* Pregnancy, planned or current
* Artificial aortic valve
* Ejection fraction less than 30 percent at baseline
* Myocardial infarction in the past 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-12; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety of treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Luis de la Fuente, MD, Principal Investigator — Argentine Institute of Diagnosis and Treatment
Locations (2):
- Argentina (2):
  - Swiss Clinic, Buenos Aires
  - Argentine Institute of Diagnosis and Treatment, Buenos Aires